CLINICAL TRIAL: NCT00003386
Title: Treatment of Ovarian Carcinoma With DNP-Modified Autologous Tumor Vaccine
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Ovarian Epithelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066382; GOG-9802
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2008-12

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — BCG Vaccine; FANG vaccine; Carboplatin; Cisplatin; Cyclophosphamide; Paclitaxel; Surgical Procedures, Operative

INTERVENTIONS:
Biological: BCG vaccine
Biological: autologous tumor cell vaccine
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: paclitaxel
Other: dinitrophenyl
Procedure: surgical procedure

SUMMARY:
RATIONALE: Vaccines made from tumor tissue may make the body build an immune response and kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have stage III or stage IV ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether patients with surgically debulked ovarian epithelial cancer develop delayed-type hypersensitivity to dinitrophenyl-modified autologous tumor vaccine. II. Assess the toxic effects of this regimen in these patients. III. Determine the feasibility of conducting a group wide vaccine study.

OUTLINE: Patients undergo a standard debulking procedure with the tumor tissue being sent to Thomas Jefferson University. Patients then receive six courses of combination chemotherapy consisting of either paclitaxel and cisplatin or paclitaxel and carboplatin. Vaccine therapy must commence within 4-12 weeks of completion of chemotherapy. Patients are tested for delayed-type hypersensitivity (DTH) on day -7. Cyclophosphamide IV is administered on day 0. Dinitrophenyl (DNP)-modified autologous ovarian epithelial cell vaccine and BCG adjuvant are injected once a week beginning on day 3 and continuing for 6 weeks. DTH testing is repeated at week 8. Booster vaccine injections are administered at 6 and 12 months if patient is disease free. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Surgically debulked stage III or IV ovarian epithelial cancer Must be able to obtain adequate number of viable cells from excised tumor mass Must have received 6 courses of combination chemotherapy comprised of either paclitaxel and cisplatin OR paclitaxel and carboplatin Must be clinically tumor free following completion of chemotherapy (i.e., no metastasis by physical examination and CT of the abdomen and pelvis and serum CA-125 less than 35 IU/L) Not on a Phase III GOG protocol

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: GOG 0 or 1 Hematopoietic: Hematocrit at least 25% WBC at least 3,000/mm3 Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing No active infections HIV negative Hepatitis B surface antigen negative Hepatitis C antibody negative No active autoimmune disease No prior invasive malignancy within the past 5 years except nonmelanomatous skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics 4-12 weeks since prior chemotherapy Endocrine therapy: No concurrent systemic corticosteroids Radiotherapy: At least 6 months since prior major field radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berd, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (60):
- United States (59):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada